CLINICAL TRIAL: NCT01992146
Title: Effect of High-dose Naloxone Infusion on Pain and Hyperalgesia in Patients Following Groin-Hernia Repair. A Randomized, Placebo-controlled, Double-blind Crossover Study
Brief Title: Effect of High-dose Naloxone Infusion on Pain and Hyperalgesia in Patients Following Groin-Hernia Repair.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: University of Kentucky (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mads Werner, Physician, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MP_SM01_2013
Record Dates: First submitted 2013-11-07; First posted 2013-11-25 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Central Nervous System Sensitization; Pain; Hyperalgesia
Keywords: central sensitization; endogenous opioids; humans; latent sensitization; naloxone; open groin hernia repair; pain; randomized controlled trial; secondary hyperalgesia; target-controlled infusion
MeSH Terms: conditions — Pain; Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Change in Pain Ratings (NRS) at the surgical site and at the mirror-site in the contralateral groin six to eight weeks after unilateral herniotomy following administration of placebo.
  Interventions: Drug: Placebo
- Target-controlled naloxone-infusion (total dose: 3.25 mg/kg) (Experimental): Change in Pain Ratings (NRS) at the surgical site and at the mirror-site in the contralateral groin six to eight weeks after unilateral herniotomy following administration of naloxone.
  Interventions: Drug: Target-controlled naloxone-infusion

INTERVENTIONS:
Drug: Target-controlled naloxone-infusion
  Arms: Target-controlled naloxone-infusion (total dose: 3.25 mg/kg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Recent studies have focused on the role of endogenous opioids on central sensitization. Central sensitization is known to be impaired or altered in chronic pain conditions, as fibromyalgia or chronic tension headache.

Animal studies have shown reinstatement of mechanical hypersensitivity following naloxone administration after resolution of an injury. This suggests latent sensitization.

In the present study, investigators hypothesize that a high-dose target-controlled naloxone infusion (total dose: 3.25 mg/kg) can reinstate pain and hyperalgesia 6-8 weeks after a unilateral primary open groin hernia repair procedure. Investigators aim to show that latent sensitization is present in humans and is modulated by endogenous opioids.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 65 years
* Signed informed consent
* Patients submitted to unilateral, primary inguinal, open herniotomy 6-8 weeks prior to study start.
* Open operating procedure a.m. Lichtenstein.
* Urin sample without traces of opioids (morphine, methadon, buprenorphine, codeine, tramadol, ketobemidone, oxycodone, hydromorphine, dextromethorphan)
* ASA I-II
* Body mass index (BMI): 18 < BMI < 30

Exclusion Criteria:

* Volunteers , who do not speak or understand Danish
* Patients, who cannot cooperate with the investigation
* Patients who have had previous surgery in the groin region
* Patients with pain at rest > 3 (NRS)
* Activity-related pain in the surgical field > 5
* Allergic reaction against morphine or other opioids (including naloxone),
* Abuse of alcohol or drugs - according to investigator's evaluation
* Use of psychotropic drugs (exception of SSRI)
* Neurologic or psychiatric disease
* Chronic pain condition
* Regular use of analgesic drugs
* Skin lesions and tattoos in the assessment areas
* Nerve lesions in the assessment sites (for instance, after trauma, disc herniation, etc.)
* Use of prescription drugs 1 week before the trial
* Use of over-the-counter drugs 48 hours before the trial

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2015-12-14 (Actual); Study Completion 2018-05-11 (Actual)

PRIMARY OUTCOMES:
Summated pain intensity | 1st session: 6-8 weeks after surgery; 2nd session: one week later
  Change in pain ratings ([NRS,0-10] pain at rest + pain during transition from supine to standing position + pain during pressure (100 kPa) at injury site), assessed 6-8 weeks after unilateral, primary, open groin hernia repair following administration of naloxone/placebo.

SECONDARY OUTCOMES:
Secondary hyperalgesia/allodynia | 1st session: 6-8 weeks after surgery; 2nd session: one week later
  Change in secondary hyperalgesia area/allodynia at surgical site and at the mirror-site in the contralateral groin assessed 6-8 weeks after unilateral, primary, open groin hernia repair following administration of naloxone/placebo.
Pressure pain thresholds | 1st session: 6-8 weeks; 2nd session: one week later
  Change in pressure pain thresholds at surgical site and at the mirror-site in the contralateral groin assessed 6-8 weeks after unilateral, primary, open groin hernia repair following administration of naloxone/placebo.

OTHER OUTCOMES:
Pain Catastrophizing Scale | in the 1st session: 6-8 weeks after surgery
  Patients fill out Pain Catastrophizing Scale before assessments on the first study day
Hospital Anxiety and Depression Scale | in the 1st session: 6-8 weeks after surgery
  Patients fill out Hospital Anxiety and Depression Scale before assessments on the first study day
Clinical Opiate Withdrawal Scale | 1st session: 6-8 weeks after surgery; 2nd session: one week later
  Clinical Opiate Withdrawal Scale is filled out before and during naloxone/placebo administration in each experimental session

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, M.D., D.M.Sc., Principal Investigator — Rigshospitalet, Denmark; Mads U Werner, M.D., D.M.Sc., Study Director — Rigshospitalet, Denmark
Locations (1):
- Multidisciplinary Pain Center, 7612, HOC, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Papathanasiou T, Springborg AD, Kongstad KT, Staerk D, Moller K, Taylor BK, Lund TM, Werner MU. High-dose naloxone, an experimental tool uncovering latent sensitisation: pharmacokinetics in humans. Br J Anaesth. 2019 Aug;123(2):e204-e214. doi: 10.1016/j.bja.2018.12.007. Epub 2019 Jan 18. PMID 30915992
- [Derived] Pereira MP, Werner MU, Dahl JB. Effect of a high-dose target-controlled naloxone infusion on pain and hyperalgesia in patients following groin hernia repair: study protocol for a randomized controlled trial. Trials. 2015 Nov 10;16:511. doi: 10.1186/s13063-015-1021-6. PMID 26554360